CLINICAL TRIAL: NCT04105270
Title: A Randomized Double Blind Phase II Trial of Restorative Microbiota Therapy (RMT) in Combination With Durvalumab (MEDI4736) and Chemotherapy in Untreated Patients With Advanced or Metastatic Adenocarcinoma Non-Small Cell Lung Cancer
Brief Title: RMT in Combination With Durvalumab + Chemo in Untreated Adenocarcinoma NSCLC. A Randomized Double Blind Phase II Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019LS010
Record Dates: First submitted 2019-09-20; First posted 2019-09-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Adenocarcinoma of Lung; Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Lung Neoplasms | interventions — Capsules; durvalumab; Cisplatin; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (RMT) (Experimental)
  Interventions: Drug: Oral Restorative Microbiota Therapy (RMT) Capsules; Drug: Durvalumab 1500 mg IV; Drug: Cisplatin/pemetrexed or Carboplatin/pemetrexed
- Arm B (Placebo) (Experimental)
  Interventions: Drug: Durvalumab 1500 mg IV; Drug: Cisplatin/pemetrexed or Carboplatin/pemetrexed; Other: Placebo
- Safety Run-in (Experimental): 10 patients are enrolled in this safety run-in arm. Patients are directly assigned to RMT treatment arm. After safety- run-in period of 4 weeks after the first dose of RMT, in the 10 patients if no new safety signal are seen enrollment moves to randomization
  Interventions: Drug: Oral Restorative Microbiota Therapy (RMT) Capsules; Drug: Durvalumab 1500 mg IV; Drug: Cisplatin/pemetrexed or Carboplatin/pemetrexed

INTERVENTIONS:
Drug: Oral Restorative Microbiota Therapy (RMT) Capsules — Patients with PD-L1 TC expression will receive sixteen doses of oral RMT capsules weekly
  Other Names: RMT
  Arms: Arm A (RMT); Safety Run-in
Drug: Durvalumab 1500 mg IV — Patients with PD-L1 TC expression receive durvalumab 1500 mg IV every 4 weeks (Q4W) until disease progression or for a maximum of two years from the 1st dose of durvalumab
Drug: Cisplatin/pemetrexed or Carboplatin/pemetrexed — Patients with PD-L1 TC receive cisplatin/pemetrexed or carboplatin/pemetrexed given every 3 weeks (Q3W) for 4 cycles followed by pemetrexed maintenance given Q3W
Other: Placebo — Sixteen doses of oral placebo capsules given weekly
  Arms: Arm B (Placebo)

SUMMARY:
This is a randomized, active-controlled, parallel-group, double-blind Phase II trial, of oral restorative microbiota therapy (RMT) or placebo combined with intravenous (IV) durvalumab (MEDI4736) plus chemotherapy in patients with treatment naïve advanced or metastatic adenocarcinoma non-small cell lung cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the lung that is unresectable stage IIIB/C or stage IV, does not have an EGFR sensitizing (activating) mutation or ALK or ROS1 translocation. BRAF, RET, NTRK, MET ex 14 splice site mutation
* Measurable disease based on RECIST 1.1
* Tumor sample requirements

  * Mandatory provision of an unstained, archived tumor tissue sample in a quantity sufficient to allow for biomarker and genomic analysis. A minimum of 10 unstained slides should be available for evaluation.
  * Known PD-L1 TC expression status assayed by Ventana SP263. Patients who have known PDL-1 as assayed by PharmDx 22C3 assay may be eligible; however, available archival tissue will be used to assay with Ventana SP263 test.
* Prior chemotherapy or immunotherapy as adjuvant therapy for lung cancer is permitted as long as it has been >6 months from last dose at the time of enrollment. Local treatment of isolated lesions, excluding target lesions, for palliative intent is acceptable (e.g. by local surgery or radiotherapy). Prior systemic therapy for advanced/metastatic NSCLC makes the patient ineligible for this study.
* Patients with treated brain metastasis are eligible as long as they have stable symptoms, are more than 2 weeks from completion of therapy, and do not require more than 10mg of daily prednisone or equivalent.
* ECOG Performance status of 0 or 1
* Body weight of >30 kg
* Adequate organ function within 14 days of study enrollment defined as:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤1.5x upper limit of normal (ULN) - this will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
  * AST (SGOT) and ALT (SGPT) ≤2.5 x institutional ULN unless liver metastases are present, in which case it must be ≤5x ULN
  * Measured creatinine clearance (CL) >40 mL/min or calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:
* Expected life expectancy of at least 12 weeks in the opinion of the enrolling investigator as documented in the medical record
* Women of childbearing potential and men with partners of child-bearing potential must agree to use effective contraception for the time of screening to the duration of treatment and 3 months after the last dose of study drug
* Provide voluntary written consent prior to the performance of any research related tests or procedures.

Exclusion Criteria:

* Not pregnant or breast feeding. Evidence of post-menopausal status, or negative urine or serum pregnancy test for female pre-menopausal patients. Women will be considered postmenopausal if they have amenorrhea for 12 months without an alternative medical explanation
* Dysphagia or inability to swallow medications
* Squamous cell, large cell, or NSCLC NOS (not otherwise specified) histology or mixed tumors
* Has untreated brain metastasis or active leptomeningeal carcinomatosis
* Has a known sensitivity to any component of therapeutic agents used in this study
* Receipt of any immunotherapy or investigational drug within 4 weeks prior to the first dose of study drug; and in the case of monoclonal antibodies 6 weeks prior to the first dose of study drug
* Prior treatment with any other anti-PD-1, or PD-L1, including durvalumab or an anti-PD-L2 agent or an antibody or a small molecule targeting other immuno-regulatory receptors except as adjuvant therapy for NSCLC so long as it has been greater than six months since the last treatment
* Current or prior use of immunosuppressive medication within 28 days before the first dose of study drug, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) that would prevent administration of study drug
* Active or prior documented autoimmune disease within the past 2 years requiring systemic treatment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Active documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis) who require immunosuppression or patients who exceed 10 mg/day of prednisone, or an equivalent corticosteroid are excluded
* History of primary immunodeficiency
* History of organ transplant that requires therapeutic immunosuppression
* Taking daily probiotics (patients with last probiotic > 4weeks prior to first dose of RMT are eligible)
* History of Human Immunodeficiency Virus (HIV) (known HIV 1/2 antibodies positive) who are on anti-retroviral treatment for < 6 months and absolute CD4 count<500 (patients with HIV not meeting these criteria are eligible)
* Has known active Hepatitis B or C. Active Hepatitis B is defined as a known positive HBsAg, and positive hepatitis B virus quantification assay (patients with history of Hepatitis B who have seroconversion i.e. Hepatitis B core antibody positive and Hepatitis B surface antibody positive are eligible). Active Hepatitis C is defined by a known positive Hep C Ab result and positive quantitative HCV RNA results (Patients with Hepatitis C who are on anti-viral suppressive therapy and negative quantitative HCV RNA results are eligible)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses
* Myocardial infarction or stroke within 3 months prior to enrollment
* History of systolic or diastolic heart failure with New York Heart Association (NYHA) class III or IV symptoms (refer to Appendix II)
* Has active or prior history of (non-infectious) pneumonitis that required steroids or patients with interstitial lung disease
* Psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent
* Known history of active tuberculosis. Patients with prior history of latent TB could be included if they have been treated previously with isoniazid.
* Patients who are on chronic systemic antibiotic therapy (antibiotics for ≥60 consecutive days within 12 weeks of enrollment). Patients who receive systemic antibiotics between enrollment and start of RMT are eligible
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving RMT
* History of another primary malignancy (excluding non-melanoma skin cancer) within 5 years prior to starting RMT, except if the patient has undergone potentially curative therapy with no evidence of disease recurrence for 5 years since initiation of that therapy
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the study drug or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing Progression Free Survival (PFS) | 3 Years
  Incidence of PFS using RECIST 1.1 in each treatment arm to evaluate the efficacy of restorative microbiota therapy
Safety and tolerability of RMT | 2 Years
  Safety and tolerability of RMT in combination with durvalumab or durvalumab + chemotherapy as assessed by the incidence of adverse events

SECONDARY OUTCOMES:
Objective Response Rate (ORR) RECIST 1.1 | 2 Years
  ORR of treatment with RMT in each treatment arm per RECIST 1.1
Duration of Response (DOR) | 2 Years
  DOR of treatment with RMT in each treatment arm per RECIST 1.1
Overall Survival (OS) | 3 Years
  Incidence of OS using RECIST 1.1 in each treatment arm
Immune mediated Adverse Events imAE | 2 Years
  Rate of immune mediated adverse events (imAE) in each treatment arm
Objective Response Rate (ORR) (iRECIST) | 2 Years
  ORR using immune response evaluation criteria in solid tumors (iRECIST)
Health-related quality of life (QoL) | 2 Years
  Difference in health-related quality of life (QoL) using European organization for research and treatment of cancer quality of life questionnaire (EORTC QLQ-30)
Health-related quality of life (QoL) | 2 Years
  Difference in health-related quality of life (QoL) using lung cancer module (LC-13)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Patel, DO, Principal Investigator — University of Minnesota, Division of Hematology, Oncology and Transplantation
Locations (10):
- United States (10):
  - Dr. Amit Kulkarni, Phoenix, Arizona
  - MNCCTN Essentia Health St. Joseph's Brainerd Medical Center, Brainerd, Minnesota
  - MNCCTN Essentia Health Deer River, Deer River, Minnesota
  - MNCCTN Essentia Health St. Mary's Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - MNCCTN Essentia Health Duluth, Duluth, Minnesota
  - MNCCTN Essentia Health Fosston, Fosston, Minnesota
  - MNCCTN Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - MNCCTN Essentia Health Sandstone, Sandstone, Minnesota
  - MNCCTN Essentia Health Virginia Clinic, Virginia, Minnesota